CLINICAL TRIAL: NCT04902872
Title: A Phase 1/2 Study of CBX-12 in Subjects With Advanced or Metastatic Refractory Solid Tumors
Brief Title: Study of CBX-12 in Subjects With Advanced or Metastatic Refractory Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cybrexa Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CBX-12-101
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumor, Adult; Epithelial Ovarian Cancer; Small Cell Lung Carcinoma; Breast Cancer; Colorectal Cancer; Pancreas Cancer; Appendix Cancer; Non-small Cell Lung Cancer; Gastric Cancer; Esophagus Cancer; Urothelial Carcinoma; Sarcoma
Keywords: SCLC; small cell lung cancer; ovarian; breast; appendix; colorectal; pancreatic; NSCLC; Sarcoma
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Small Cell Lung Carcinoma; Breast Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Appendiceal Neoplasms; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Esophageal Neoplasms; Carcinoma, Transitional Cell; Sarcoma

STUDY DESIGN:
Intervention Model Description: Parts B, C & Modified Part B will follow a 3 + 3 design, enrolling 3 subjects in each cohort. (De)escalation rules: DLT period for each subject in Phase 1 Part B & Modified Part B will be 3 weeks & 4 weeks in Part C (i.e., 1 cycle). If none of the 3 subjects experience a DLT, dose will be escalated to next highest dose level. If 1 of 3 subjects in cohort experiences a DLT, up to 3 additional subjects will be enrolled/treated at same dose. If none of the additional 3 subjects experience a DLT (i.e., only 1 of 6 subjects in cohort has a DLT), dose will be escalated to next highest level. If 2 or more of up to 6 subjects at dose level have DLTs, enrollment to that cohort will stop, dose will be considered above MTD. Dose will be decreased to previous dose level or to a level intermediate to those previously evaluated. MTD will be highest dose evaluated at which ≤ 1 of 6 have a DLT. A minimum of 6 DLT-evaluable subjects will be enrolled to any dose level being evaluated as possible MTD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Phase 1 Schedule B Dose Escalation (Daily Dosing x 3) (Experimental): CBX-12 administered on a daily x 3, 3 week schedule
  Interventions: Drug: CBX-12
- Phase 1 Schedule C Dose Escalation (Once Weekly Dosing ) (Experimental): CBX-12 administered once weekly, 4 week schedule
  Interventions: Drug: CBX-12
- Phase 2 Ovarian Cancer Expansion Cohort (Experimental): CBX-12 administered TBD
  Interventions: Drug: CBX-12
- Phase 2 Metastatic Breast Expansion Cohort (Experimental): CBX-12 administered TBD
  Interventions: Drug: CBX-12
- Phase 1 Schedule A Dose Escalation (Daily Dosing x 5) (Experimental): CBX-12 administered on a daily x 5, 3 week schedule
  Interventions: Drug: CBX-12
- Phase 1 Modified Schedule B Dose Escalation (Once Every 3 weeks) (Experimental): CBX-12 administered once every 3 weeks
  Interventions: Drug: CBX-12

INTERVENTIONS:
Drug: CBX-12 — CBX-12 is an alphalex construct which consists of a low-pH insertion peptide, a self-immolating linker, and exatecan as the pharmacologically active moiety

SUMMARY:
This is a first-in-human, Phase 1/2 open-label, multicenter, dose-escalation, safety, pharmacokinetics (PK), and biomarker study of CBX-12 in subjects with advanced or metastatic refractory solid tumors.

DETAILED DESCRIPTION:
Phase 1 is the dose-escalation portion of the study in which the safety and tolerability of three dosing schedules of CBX-12 will be evaluated. Subjects in Part A will be treated with CBX-12 on a daily x 5 every 3 weeks schedule (treatment in Part A was discontinued in October 2021). Subjects in Phase 1 Part B will be treated with CBX-12 on a daily x 3 every 3 weeks schedule. Subjects in Phase 1 Part C will be treated with CBX-12 once weekly. Subjects in Phase 1 Modified Part B will be treated with CBX-12 once every 3 weeks.

For all parts in Phase 1, after all subjects in a cohort have completed treatment through the DLT period or discontinued treatment due to a DLT, the SRC, composed of the Investigators who have enrolled subjects in the current cohort(s), the study Medical Monitor and ad hoc members (e.g., other Investigators, a statistician) as needed, will review all available safety data, including DLTs and all available PK data for that cohort and make dose-level recommendations.

Once the recommended phase 2 dose (RP2D) has been established in Part B, Part C and Modified Part B, Phase 2 expansion cohorts may open.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject has a histologically- or cytologically-diagnosed solid tumor which is advanced or metastatic and which has progressed on or following at least one systemic therapy regimen administered for advanced or metastatic disease or for which no approved therapy exists. Subject's prior treatment should include all approved regimens that have demonstrated a survival advantage for the subject's disease, stage, and line of therapy.
* Has measurable disease per RECIST 1.1.
* An adequate tumor sample must be available from core needle biopsies obtained during the Screening Period and following the subject's most recent systemic therapy.
* Agrees to an on-treatment biopsy preferably of the same lesion from which the pre-CBX-12 treatment sample was obtained as long as the Investigator determines such biopsy can be performed with acceptable safety. (Removed Amd 4, date 31-Mar-2023)

Exclusion Criteria:

* Cytotoxic chemotherapy, biologic agent, investigational agent, or radiation therapy less than or equal to 3 weeks prior to the first dose of CBX-12. The interval may be reduced to 2 weeks for bone only radiation therapy or investigational agents not expected to be associated with adverse events (AEs) after 2 weeks of last administration, with Medical Monitor approval.
* Small-molecule kinase inhibitors or hormonal agents less than or equal to 14 days prior to the first dose of CBX-12.
* Subjects who are currently receiving any other anti cancer or investigational agent(s).
* Clinically significant intercurrent disease.
* Subjects with primary central nervous system (CNS) tumors or clinically active CNS metastases or carcinomatous meningitis. Subjects with stable brain metastasis may be enrolled with Medical Monitor approval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of treatment-emergent adverse events (TEAEs) | Through the end of study, estimated as 6 months
  NCI CTCAE v5.0
Phase 1: Recommended Phase 2 Dose for Daily x 3 every 3 weeks schedule of CBX-12 (Schedule B) | 15 months
  Safety Review Committee Analysis of Safety and PK Data
Phase 1: Recommended Phase 2 Dose for Once Weekly schedule of CBX-12 (Schedule C) | 15 months
  Safety Review Committee Analysis of Safety and PK Data
Phase 1: Recommended Phase 2 Dose for Once Every 3 Weeks schedule of CBX-12 (Modified Schedule B) | 15 months
  Safety Review Committee Analysis of Safety and PK Data
Phase 2: Overall response rate (ORR) | Through the end of study, estimated as 6 months
  ORR Based on RECIST v1.1

SECONDARY OUTCOMES:
Maximum concentration of CBX-12 | 5 days
  PK Analysis
Area under the curve from 0-24 hours of CBX-12 | 5 days
  PK Analysis
Time to maximum concentration of CBX-12 | 5 days
  PK Analysis
Half-life of CBX-12 | 5 days
  PK Analysis
Clearance (CL) of CBX-12 | 5 days
  PK Analysis
Apparent Volume of Distribution at Steady State (Vss) CBX-12 | 5 days
  PK Analysis
Phase 1: ORR | Through the end of study, estimated as 6 months
  Based on RECIST v1.1
Duration of Response (DoR) | Through the end of study, estimated as 6 months
  Based on RECIST v1.1
Progression-free Survival (PFS) | Through the end of study, estimated as 6 months
  Based on RECIST v1.1
Phase 2: Incidence of TEAEs | Through the end of study, estimated as 6 months
  NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Yale Cancer Center, New Haven, Connecticut
  - NEXT Oncology, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No